CLINICAL TRIAL: NCT04036123
Title: Assessment of the Lower Urinary Tract: Consistency, Features and Artifacts of Invasive Urodynamic Assessments - Synchrony
Brief Title: Urodynamic Assessment of the Lower Urinary Tract: Water vs. Air - Synchrony
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UDI-Synchrony 2018-00073
Record Dates: First submitted 2019-07-19; First posted 2019-07-29 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Lower Urinary Tract Dysfunction
Keywords: Urodynamic investigation; Lower urinary tract dysfunction; Water-perfused catheter; Air-charged catheter

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Urodynamic investigation (Experimental): Simultaneous UDI (same session repeat filling cystometry and pressure flow study) with an air-charged and water-perfused measurement system.
  Interventions: Other: Urodynamic investigation

INTERVENTIONS:
Other: Urodynamic investigation — Simultaneous UDI (same session repeat filling cystometry and pressure flow study) with an air-charged and water-perfused measurement system.

SUMMARY:
Comparison of water-perfused (WP) and air-charged (AC) catheters for invasive urodynamic investigation (UDI) regarding consistency, features and artifacts.

DETAILED DESCRIPTION:
UDI is the gold standard to assess refractory lower urinary tract symptoms (LUTS), i.e. to detect and specify lower urinary tract dysfunction (LUTD). Therefore, UDI findings lead to diagnosis and decision-making for further non-invasive and invasive therapies. For UDI pressure recordings, the use of WP catheters is recommended by the International Continence Society (ICS).

Currently AC catheters have been marked for pressure recording as an alternative to WP catheters. However, the number of comparative studies is very limited. Nevertheless, since release, AC catheters have gained popularity due to their omnidirectional detection of pressure, and claimed reduction in movement artefacts (due to weight-less air column vs weighted water column), lack of external reference level, and ease of set-up/use. Still, there is debate whether AC catheters are an acceptable alternative to fluid-filled lines for measuring intravesical and intra-abdominal pressure in UDI. Based on the available literature, an appropriate conclusion, whether both systems can be used as equivalents and interchangeably, cannot be drawn.

In this study, the investigators compare both systems regarding consistency, features and artifacts.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Age ≥18 years
* Informed consent
* LUTD due to a neurological disorder
* Competent German language skills

Exclusion Criteria:

* Age <18 years
* Pregnancy or breast feeding (see chapter 3.6.)
* Symptomatic UTI
* Individuals especially in need of protection
* No informed consent
* Patients incapable to follow the trial, e.g. because of language problems, psychiatric disorders, dementia and so on.
* Earlier participation in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Interchangeability of the measurement method (air-charged vs. water-perfused measurement system) regarding the urodynamic observations, diagnostic result and subsequent treatment | Once during urodynamic investigation

SECONDARY OUTCOMES:
Pressure changes during urodynamics using an air-charged vs. water-perfused measurement system | Once during urodynamic investigation
  Maximum DO amplitude [cmH2O], detrusor leak-point pressure [cmH2O], maximum detrusor pressure [cmH2O] during storage phase, maximum detrusor pressure [cmH2O] during voiding phase, detrusor pressure at maximum flow rate [cmH2O]
Changes in bladder compliance [mL/cmH2O] during urodynamics using an air-charged vs. water-perfused measurement system | Once during urodynamic investigation]
Incidence of side effects: number and intensity/severity (mild/moderate/severe) of AEs and SAE for the following categories during and for 7 days after the urodynamic investigation | Once during urodynamic investigation and 7 days thereafter
  Infection - Urinary Tract Infection (UTI); severe or sudden increase in pain; severe or sudden increase in spasticity; autonomic dysreflexia; urgent (unexpected) transfer/admittance to an acute care facility

CONTACTS AND LOCATIONS:
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland